CLINICAL TRIAL: NCT00117533
Title: A Pilot Study to Evaluate the Efficacy and Safety of Pegylated Interferon Alfa-2b Plus Ribavirin in the Treatment of Patients With Dual Chronic Hepatitis B and Delta
Brief Title: Pegylated Interferon Alfa-2b Plus Ribavirin in Chronic Hepatitis B and Delta
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); National Science and Technology Council, Taiwan (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 930904
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2006-05-25 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis B; Chronic Hepatitis D
Keywords: chronic hepatitis B;; chronic hepatitis delta;; treatment;; pegylated interferon alfa-2b;; ribavirin
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis D, Chronic | interventions — Ribavirin

INTERVENTIONS:
Drug: pegylated IFN alfa-2b plus ribavirin

SUMMARY:
The treatment of choice for chronic hepatitis D is uncertain. The investigators hypothesize that pegylated interferon (IFN) alfa-2b in combination with ribavirin (RBV) may be effective in the treatment of chronic hepatitis D patients who are also infected by hepatitis B virus (HBV). The purpose of this study is to test this hypothesis. The investigators will use pegylated IFN alfa-2b in combination with RBV for the treatment of patients with dual chronic hepatitis D virus (HDV) and HBV infection. A 24-week course of combination therapy pegylated IFN+RBV will be used.

DETAILED DESCRIPTION:
Recombinant IFN alfa possesses anti-viral and immunomodulatory effects and has been shown to be effective in chronic hepatitis B [Davis et al. 1989; Bisceclie et al, 1989]. Interferon alfa is also one of the approved treatments for chronic hepatitis B. Administration of IFN alfa-2b to adults leads to disappearance of HBV DNA with or without HBeAg seroconversion in 30-50% of patients, which is two to three times above the rate of yearly spontaneous HBeAg seroconversion (10-15%). Normalization of serum ALT occurs in most cases. Loss of HBsAg is observed in 10-15% of Caucasian patients during the prolonged post-treatment follow-up period. Recently, studies suggested that a higher proportion of patients receiving pegylated IFN could achieve HBeAg seroconversion and control of HBV replication [Marcellin et al, 2004; Lau et al, 2004; Jensen et al, 2004].

RBV is another antiviral nucleotide analogue with few adverse effects [Sidwell et al, 1972; Patterson et al, 1990]. RBV alone can modestly inhibit HDV or HBV replication [Choi et al, 1989]. The beneficial effect of combined IFN plus RBV in the treatment of chronic hepatitis B has also been shown in previous studies [Cotonat et al, 2000]. Why RBV can greatly enhance the treatment efficacy is not clear. It had been shown that ribavirin could inhibit interleukin-4, an inhibitor of cytotoxic T lymphocyte activity, and preserves the interleukin-2 and gamma IFN activities. Other studies revealed that the enhanced efficacy was associated with HBV- or other virus-specific type 1 cytokine-mediated T helper cell responses [Cramp et al, 2000; Tam et al, 1999; Hultgren et al, 1998; Fang et al, 2002; Fang et al, 2000; Rico et al, 2001]. Thus, the combination therapy may augment virus-specific cytotoxic T lymphocytes and non-specific immune response, and effectively shift the immune responses to the more potent antiviral type 1 T-helper profile [Hultgren et al, 1998].

HDV, like HCV, is a RNA virus. Indeed, RBV had also been shown to be active against HDV replication in cell cultures [Choi et al, 1989]. The investigators therefore hypothesize that pegylated IFN alfa-2b in combination with RBV can yield an efficacy in chronic hepatitis D patients who are dually infected by HBV. The purpose of this protocol is to test this hypothesis. A previous study found that high-dose IFN may improve the efficacy for chronic hepatitis D patients. Another pilot study using IFN alfa plus RBV also demonstrated that the seroclearance of HCV RNA was not affected by HBV coinfection [Liu et al, 2003]. The investigators thus use pegylated IFN alfa-2b in combination with RBV for the treatment of patients with dual chronic HDV and HBV infection.

The treatment choice for chronic hepatitis D was not clarified till now. In this proposal, the dosage and duration for the combination regimen are decided mainly by the experience from the treatment of chronic hepatitis B and chronic hepatitis C.

The investigators recent study using ribavirin and interferon (IFN) combination therapy for dual chronic hepatitis B and C suggested that combining ribavirin 1,200 mg daily for 6 months, together with 6 million units (MU) IFN-alpha 2a thrice weekly for 12 weeks and then 3 MU for another 12 weeks was effective for the clearance of HCV RNA [Liu et al, 2003]. Twenty-four patients with chronic hepatitis seropositive for both hepatitis B surface antigen and antibody to HCV received ribavirin 1,200 mg daily for 6 months, together with 6 million units (MU) IFN-alpha 2a thrice weekly for 12 weeks and then 3 MU for another 12 weeks. The serum HCV clearance rate was 43% 24 weeks posttreatment. The serum ALT normalization rate was 43% 24 weeks posttreatment. In hepatitis B and C dually infected patients, combination IFN with ribavirin can achieve a sustained HCV clearance rate comparable with hepatitis C alone. Furthermore, a previous study revealed that a 12-week RBV therapy was not effective for patients with chronic hepatitis B [Kakumu et al, 1993]. Therefore, a 24-week course of combination therapy pegylated IFN+RBV will be used.

Increased RBV dosage has been considered a contributory factor to the better efficacy in treating refractory genotype HCV. For example, recent studies suggested that using RBV 800 mg daily is adequate to treat HCV genotype non-1 while the standard dosage of RBV is required to treat HCV genotype 1 [NIH 2002]. The investigators thus propose to use RBV 1000-1200 mg daily according to the body weight of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Be positive for both anti-HDV and HBsAg for more than 6 months
* Present with elevated serum ALT levels at least 1.5 times the upper limit of normal, documented on two occasions (at least one month apart), within six months prior to enrollment
* Be HDV RNA positive by PCR (sensitivity: 103 copies/mL) [Yamashiro et al, 2004]
* Be HBV DNA positive by PCR
* Present with liver biopsy findings compatible with the diagnosis of chronic liver disease (the liver biopsy needs to be taken within 52 weeks prior to enrollment)
* Have adequate liver reserve (defined as equal to or better than Child-Pugh Class A)
* Present with WBC ≥3000/mm3, ANC ≥1500/mm3, and platelet ≥80,000/mm3
* Be able to and likely to attend regularly for treatment and follow-up
* Give their written informed consent
* Be negative for urine pregnancy test (for females of childbearing potential), documented once within the screening period and again within 24 hours prior to the first dose of study drug
* All male patients with female partners of childbearing age should use a barrier method of contraception
* All female patients of childbearing potential must use two reliable forms of effective contraception

Exclusion Criteria:

* Drug addicts or have any history or histological evidence of alcohol abuse, or currently receive prescriptions that may cause hepatotoxicity
* Have decompensated cirrhosis as coded by Child-Pugh classification (i.e. history of ascites, history of bleeding from esophageal varices, severe portal hypertension, serum albumin <30 g/l, serum bilirubin >30 mg/l)
* Present with WBC <3000/mm3, ANC <1500/mm3, or platelets <90,000/mm3
* Present with hemoglobin <12.0 gm/dl for female and <13.0 gm/dl for male
* Have been treated with immunosuppressive therapy within the past six months (e.g. steroids, azathioprine, cyclophosphamide)
* Have renal insufficiency (serum creatinine >150 μmol/l)
* Have clotting abnormalities which preclude a liver biopsy
* Have evidence of any serious neurological dysfunction
* Have obesity or diabetes mellitus-induced liver disease
* Have serological evidence of autoimmune chronic liver disease (e.g. antinuclear antibody titers >1:320, and/or smooth muscle antibody titers>1:160)
* Hemophiliacs
* Have evidence of inheritable disorders such as haemochromatosis, alpha-1-antitrypsin deficiency or Wilson's disease
* Have been exposed to hepatotoxic substances which might be the cause of hepatitis
* Pregnant, lactating or not practicing an adequate form of birth control, such as oral contraceptives or intrauterine devices
* Seropositive for anti-HIV or anti-HCV
* Have serious psychological or psychiatric problems disrupting daily activities
* Have AFP (alpha-fetoprotein) greater than 20 ng/ml; in case of elevated AFP, abdomen ultrasonography is required to exclude the possibility of HCC
* Have serious heart diseases (coronary heart disease, etc)
* Have a history of asthma or drug allergy which may lead to hypersensitivity to ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-09; Study Completion 2007-06

PRIMARY OUTCOMES:
the efficacy of 24-week pegylated IFN alfa-2b plus RBV for SVR of HDV in patients with dual chronic hepatitis D and B

SECONDARY OUTCOMES:
the efficacy of pegylated IFN alfa-2b plus RBV in patients with dual chronic hepatitis D and B on: The biochemical response rate
The degree of histologic change

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taipei
  - National Taiwan University, Taipei, Taipei